CLINICAL TRIAL: NCT03941041
Title: Impact of Prenatal Yoga Practice on Birth Outcome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Maribor (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRP-2018-3
Record Dates: First submitted 2019-03-21; First posted 2019-05-07 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Pregnancy
Keywords: Yoga; Caesarean Section; Delivery Outcome; Labour Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prenatal Yoga Practice (Experimental): Pregnant women participating in a yoga course at least 12 session, each session in duration of 90 minutes.
  Interventions: Behavioral: Prenatal Yoga Course
- Regular Prenatal Care (No Intervention): Pregnant women being treated according to national guidelines

INTERVENTIONS:
Behavioral: Prenatal Yoga Course — participation in a 12-week prenatal yoga course (optimally), 1 session in duration of 90 minutes per week
  Arms: Prenatal Yoga Practice

SUMMARY:
Yoga is a body-mind practice that encompasses a system of postures (asana), stretching exercises combined with breathing (pranayama) and meditation (dharana). About 70% of practitioners are women, the majority of them in their reproductive age. Yoga is on the rise among pregnant women. Prenatal yoga appears to help pregnant women develop mental and physical health and build a connection with their unborn baby. It reduces stress and anxiety, lower back pain, carpal tunnel syndrome symptoms, nausea, headaches and shortness of breath, improves sleep and increase strength, flexibility and endurance of muscles needed for childbirth. A limited number of prospective randomized trials exist about the benefits of yoga in pregnancy and childbirth. An analysis of how yoga exercises in pregnancy affect the labour pattern, the outcome as well as the caesarean rate in a population of European pregnant women will be performed.

DETAILED DESCRIPTION:
Detailed Description:

The study will be a single-blind, prospective, randomised, controlled, clinical trial, with parallel assignment. Investigators intent to analyse labour patterns and outcomes in population of pregnant women which will be divided in a group that will practice yoga and a group that will not. Study will take place at the Department for Perinatology, University Medical Centre Maribor in Slovenia, Central Europe. Both groups will receive standard prenatal care. The intervention group will attend yoga classes 3 times a month. Yoga intervention will be strictly designed, lasting 90 minutes, starting at 12-14 weeks of gestation till delivery. Both groups are intended to give birth at the Department of Perinatology, University Medical Centre Maribor, Slovenia, where we have around 2200 deliveries per year.

Maribor is a university and metropolitan city as well as an educational, cultural, administrative, economic, financial, commercial and tourist centre of the north-eastern part of Slovenia with around 95.000 inhabitants.

Recruitment process Participants will be informed about the study at their gynaecologist at primary health care level in Maribor, Slovenia. Primary level gynaecologists will direct participants. Women at 12-14th week of gestation will approach the research stuff at the reception of Department of Perinatology, University Medical Centre Maribor. Participants will be introduced to the project Yoga in pregnancy. Then they will be escorted by the staff to a private room, where the study will be explained in details. Participants will be screened using written protocol. Qualified pregnant women will have the opportunity to sign a informed consent. When the informed consent is signed, the recruitment process will be completed.

Randomization Investigators will use simple randomisation of pregnant women in two groups: yoga and control. The selection (yoga or control) will be printed and placed in opaque envelopes, which will be kept and locked in a cabinet. Recruited pregnant women will be given an ID code and permit to pick one of the available envelopes to determine the group selection.

Blinding The outcome assessors will be blind for group selection: the physicians, midwifes, nurses and hospital staff.

Intervention The yoga group will receive standard care, plus yoga intervention on average 3 times a month lasting 90 minutes, beginning at 12 -14th week of gestation to the end of pregnancy. The goal is that a woman completes 12 sessions. The control group will receive standard prenatal care. The yoga practice will be conducted according to yoga system of the author Swami Maheshwarananda, named "Yoga in Daily Life" by well - trained, certified yoga teacher. Standard care for both groups include regular check-ups by the gynaecologists.

Four categories of yoga intervention will be offered to the study group:

deep relaxation practice, yogic postures, breathing exercises, meditation and visualisation exercises. Longer relaxation: 7-10 minutes, lying postures on the left side of the body is performed in the beginning of the practice. Two shorter relaxation exercises lasting 2-3 minutes are performed between yogic postures and at the beginning of the meditation and visualisation. Yoga postures will strengthen the body core and pelvic floor muscles. Meditative exercises include visualization, guided imagery and sound resonance techniques that supports the emotional bonding with the unborn baby. Participants will be asked to visualize the fetus in the uterus, the umbilical cord and the placenta. Then they will be guided to imagine the blood flow from their bodies into the placenta, through the umbilical cord, and bring nourishment, accompanied by positive emotions to their fetuses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women nulliparous women with singleton pregnancy included in the study during 12-14th week of pregnancy
* Body Mass Index between 18-30 kg/m2
* Height above 160 cm
* normal pelvic measurements (distantia spinarum: 24-26 cm; diastantia cristarum: 26-28 cm; diastantia trochanterica: 28-30 cm)
* without known anomalies of the fetus
* regular antenatal check-ups
* yoga naive

Exclusion Criteria:

* multiple pregnancy (twins, triplets ...)
* contraindications for physical activity in pregnancy (vaginal bleeding, cervical insufficiency, cerclage, placenta praevia)
* chronic diseases of the pregnant patient (hypertension, diabetes, diseases of the heart of lungs, hematological diseases)
* anomalies of the reproductive tract
* previous experience with yoga courses prior to pregnancy

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of caesarean section | Through study completion, an average 1 year
  yes/no
Rate of spontaneous vaginal birth | Through study completion, an average 1 year
  yes/no

SECONDARY OUTCOMES:
The level of pain at the 1st stage of labour | The pain is assessed before pain management in the delivery ward. Assessment through VAS (Visual Analogue Scale:1-10; in wich 1 represent no pain and 10 most severe pain participants had ever experienced).
  The pain is assessed before pain management in the delivery ward. Assessment through VAS (Visual Analogue Scale).
Rates of requests for epidural analgesia | Requests at time of admission to delivery ward
  yes/no
The assesment of anxiety in pregnancy and prior to delivery | First measurements between 12th and 14th week of pregnancy, second measurement between 36th and 38th week
  Using the STAI - State-Trait Anxiety Inventory. The study will use both, STAI-X1 and STAI-X2. STAI-X1 assesses current states of anxiety and STAI-X2 assesses anxiety as a personality trait. The Likert scale consist of 4 possible answers for statements assessing anxiety (ranging from never to very). According to the answers a key for evaluation is provided.
The assessment of childbirth anxiety (W-DEQ - The Wijma Delivery Expectancy/Experience Questionnaire) | First measurements between 12th and 14th week of pregnancy, second measurement between 36th and 38th week
  W-DEQ A questionnaire have 33 items. Woman is instructed to rate her personal feelings and cognitions on a six-point Likert scale with the endpoints market with "not at all" and "extremely" (0-5). The minimum score is 0, and the maximum score 165. The higher the score, the greater the fear of childbirth manifested.
The locally validated locally Pregnancy Concerns Scale (LJZT) Questionnaire of anxiety in pregnancy | First measurements between 12th and 14th week of pregnancy, second measurement between 36th and 38th week
  PCS have 16 items. Participant rate her personal feelings on a four-point scale with endpoints "not concerned" and "pronounced concerned" (0-3). The minimum score is 0, and the maximum score 48.

CONTACTS AND LOCATIONS:
Overall Officials: Lucija Kuder, MD, Principal Investigator — UMC Maribor; Vesna Elvedi Gasparovic, MD, PhD, Study Chair — Clinical Hospital Centre Zagreb; Faris Mujezinovic, MD, PhD, Study Chair — UMC Maribor
Locations (1):
- University Medical Center Maribor, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Babbar S, Shyken J. Yoga in Pregnancy. Clin Obstet Gynecol. 2016 Sep;59(3):600-12. doi: 10.1097/GRF.0000000000000210. PMID 27152528
- [Background] Jiang Q, Wu Z, Zhou L, Dunlop J, Chen P. Effects of yoga intervention during pregnancy: a review for current status. Am J Perinatol. 2015 May;32(6):503-14. doi: 10.1055/s-0034-1396701. Epub 2014 Dec 23. PMID 25535930
- [Background] Chuntharapat S, Petpichetchian W, Hatthakit U. Yoga during pregnancy: effects on maternal comfort, labor pain and birth outcomes. Complement Ther Clin Pract. 2008 May;14(2):105-15. doi: 10.1016/j.ctcp.2007.12.007. Epub 2008 Mar 4. PMID 18396254
- [Background] Babbar S, Hill JB, Williams KB, Pinon M, Chauhan SP, Maulik D. Acute feTal behavioral Response to prenatal Yoga: a single, blinded, randomized controlled trial (TRY yoga). Am J Obstet Gynecol. 2016 Mar;214(3):399.e1-8. doi: 10.1016/j.ajog.2015.12.032. Epub 2015 Dec 22. PMID 26721782
- [Background] Jahdi F, Sheikhan F, Haghani H, Sharifi B, Ghaseminejad A, Khodarahmian M, Rouhana N. Yoga during pregnancy: The effects on labor pain and delivery outcomes (A randomized controlled trial). Complement Ther Clin Pract. 2017 May;27:1-4. doi: 10.1016/j.ctcp.2016.12.002. Epub 2016 Dec 23. PMID 28438273